CLINICAL TRIAL: NCT03979885
Title: Financial Incentives for Smoking Treatment
Brief Title: Financial Incentives for Smoking Treatment II
Acronym: FIESTA II
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: NYU Langone Health (Other); Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Principal Investigator, Soma Wali, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA045688-01A1 (NIH)
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Smoking Cessation; Tobacco Use Cessation
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Goal-Directed Incentives (Other)
  Interventions: Behavioral: Smoking cessation counseling (Quitline); Behavioral: Smoking cessation pharmacotherapy (e.g, nicotine replacement therapy); Behavioral: Financial incentives for use of evidence-based smoking cessation therapies
- Outcome-Based Incentives (Other)
  Interventions: Behavioral: Smoking cessation counseling (Quitline); Behavioral: Smoking cessation pharmacotherapy (e.g, nicotine replacement therapy); Behavioral: Financial incentives for smoking cessation
- Enhanced Usual Care (Other)
  Interventions: Behavioral: Smoking cessation counseling (Quitline); Behavioral: Smoking cessation pharmacotherapy (e.g, nicotine replacement therapy)

INTERVENTIONS:
Behavioral: Smoking cessation counseling (Quitline) — Quitline offers community-based counseling session with a cessation counselor.
Behavioral: Smoking cessation pharmacotherapy (e.g, nicotine replacement therapy) — Participants will be encouraged to speak to their doctors about using highly effective pharmacotherapies for smoking cessation.
Behavioral: Financial incentives for smoking cessation — Participants will receive financial incentives for bioconfirmed smoking cessation.
  Arms: Outcome-Based Incentives
Behavioral: Financial incentives for use of evidence-based smoking cessation therapies — Participants will receive financial incentives for the use of evidence-based smoking cessation therapies including Quitline counseling, community-based smoking cessation programs and pharmacotherapies
  Arms: Goal-Directed Incentives

SUMMARY:
Financial incentives for motivating changes in health behavior, particularly for smoking and other morbid habits, are increasingly being tested by health insurers, employers, and government agencies. However, in using incentive programs for smoking cessation, key unanswered structural and theoretical questions remain regarding their effectiveness, acceptability to patients, and economic sustainability. This trial aims to advance the science and implementation of financial incentives for smoking cessation interventions among high-risk, hospitalized smokers. The investigators will pursue two specific aims: 1) comparing the impact of three approaches for smoking cessation on smoking abstinence, use of evidenced-based therapy, and quality of life and 2) comparing the short-term and long term return on investment of using goal directed and outcome-based financial incentives to promote smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years
2. smoked tobacco during the prior 30 days,
3. have an active U.S. phone number and address,
4. can provide consent in English or Spanish and
5. are in at least the contemplative stage of change for quitting smoking, as assessed by a single measure, readiness to quit

Exclusion Criteria:

1. use only smokeless tobacco,
2. are pregnant or breastfeeding,
3. are discharged to an institution (e.g., nursing home, long-term care facility),
4. are unable to provide informed consent, or do not have cognitive ability to enroll or participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1058 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence assessed by self-report and biochemically verified by salivary cotinine | 6 months
  Assessed by self-report questionnaire, and biochemically verified by salivary cotinine

SECONDARY OUTCOMES:
Use of evidence based treatment (e.g. counseling and smoking cessation medications) assessed by discharge prescriptions, Quitline records, receipts, letters and/or self-report | 2 months
  Assessed by discharge prescriptions, Quitline records, receipts, letters and/or self-report
Quality of life as measured by PROMIS-29 Profile v2.0 | 12 months
  Assessed by phone interviews.
Short term return on investment of using financial incentives to promote smoking cessation (Cost analysis) | 12 months
  Cost analysis involving hospital utilization data, electronic health records and patient-reported healthcare utilization
Long term return on investment of using financial incentives to promote smoking cessation (Cost analysis) | 3 years
  Cost analysis involving hospital utilization data, electronic health records and patient-reported healthcare utilization

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ladapo, MD, PhD, Principal Investigator — University of California, Los Angeles; Scott Sherman, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - David Geffen School of Medicine, Los Angeles, California
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
UCLA is committed to the ideals of collaborative research and adheres to the sponsors Grant Policy on Sharing of Unique Research Resources. Requests for research resources generated as part of this project will be distributed in a timely manner.
  Publication of data shall occur during or at the end of the project, consistent with normal scientific practices. Research data that documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Data will be redacted to prevent the disclosure of personal identifiers.

REFERENCES:
- [Derived] Wali S, Gaitonde A, Sherman S, Min N, Pesantes A, Bidgoli A, Shirley A, Tseng CH, Ladapo J. Goal-directed versus outcome-based financial incentives for smoking cessation among low-income, hospitalised patients: rationale and design of the Financial Incentives for Smoking Treatment II (FIESTA II) randomised controlled trial. BMJ Open. 2023 Sep 29;13(9):e074354. doi: 10.1136/bmjopen-2023-074354. PMID 37775282